CLINICAL TRIAL: NCT02854631
Title: A Phase 2, Double-Blind, Randomized Study Evaluating the Safety, Tolerability, and Efficacy of GS-4997 in Combination With Prednisolone Versus Prednisolone Alone in Subjects With Severe Alcoholic Hepatitis (AH)
Brief Title: Selonsertib in Combination With Prednisolone Versus Prednisolone Alone in Participants With Severe Alcoholic Hepatitis (AH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-416-2124; 2016-000821-37 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Alcoholic Hepatitis (AH)
Keywords: Cirrhosis; Prednisone; Jaundice
MeSH Terms: conditions — Hepatitis, Alcoholic; Fibrosis; Jaundice | interventions — selonsertib; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selonsertib + Prednisolone (Experimental): Selonsertib + prednisolone for 28 days
  Interventions: Drug: Selonsertib; Drug: Prednisolone
- Prednisolone (Placebo Comparator): Selonsertib placebo + prednisolone for 28 days
  Interventions: Drug: Prednisolone; Drug: Placebo

INTERVENTIONS:
Drug: Selonsertib — 18 mg tablet administered orally once daily
  Other Names: GS-4997
  Arms: Selonsertib + Prednisolone
Drug: Prednisolone — 40 mg (4 x 10 mg tablets) administered orally once daily
Drug: Placebo — Selonsertib placebo tablet administered orally once daily
  Arms: Prednisolone

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of selonsertib (GS-4997) in combination with prednisolone versus prednisolone alone in participants with severe alcoholic hepatitis (AH).

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to give informed consent prior to any study specific procedures being performed. In individuals with hepatic encephalopathy (HE) which may impair decision-making, consent will be obtained per hospital procedures (eg, by Legally Authorized Representative)
* Clinical diagnosis of severe AH

  * Maddrey's Discriminant Function (DF) ≥ 32 at screening

Key Exclusion Criteria:

* Pregnant or lactating females;
* Other causes of liver disease including chronic hepatitis B (hepatitis B surface antigen [HBsAg] positive), chronic hepatitis C (HCV RNA positive), acetaminophen hepatotoxicity, biliary obstruction, and autoimmune liver disease;
* Serum aspartate aminotransferase (AST) >400 U/L or alanine aminotransferase (ALT) >300 U/L;
* Model for End Stage Liver Disease (MELD) >30 at screening;
* Maddrey's DF >60 at screening;
* Grade 4 Hepatic Encephalopathy (HE) by West Haven criteria;
* Concomitant or previous history of hepatocellular carcinoma;
* History of liver transplantation;
* HIV Ab positive;
* Clinical suspicion of pneumonia;
* Uncontrolled sepsis;
* Uncontrolled gastrointestinal (GI) bleeding or controlled GI bleeding within 7 days of screening that was associated with shock or required transfusion of more than 3 units of blood;
* Type 1 hepatorenal syndrome (HRS) or renal failure defined as a serum creatinine >221 μmol/L (>2.5 mg/dL) or the requirement for renal replacement therapy;
* Individuals dependent on inotropic (eg, epinephrine or norepinephrine) or ventilatory support (ie, endotracheal intubation or positive-pressure ventilation);
* Portal vein thrombosis;
* Acute pancreatitis;
* Cessation of alcohol consumption for more than 2 months before Baseline/ Day 1

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (44):
- United States (11):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Research Centers, Coronado, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Cleveland Clinic Florida, Weston, Florida
  - Oschner Medical Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Methodist Healthcare Dallas - The Liver Institute, Dallas, Texas
  - Liver Institute of Virginia, Newport News, Virginia
  - University of Washington, Seattle, Washington
- Austria (3):
  - Medizinische Universitat Graz, Graz
  - Universitätsklinik für Innere Medizin I, Innsbruck
  - Medical University Vienna, Vienna
- Belgium (5):
  - Cliniques Universitaires UCL Saint-Luc, Brussels
  - CUB Hopital Erasme, Brussels
  - Ghent University Hospital, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Toronto General Hospital, Toronto, Ontario
- France (10):
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - Hôpital Jean Minjoz, Besançon
  - C.H.U. de Caen, Caen
  - CHU henri Mondor, Créteil
  - CHU de Grenoble- Hopital Michallon, La Tronche
  - CHRU de Lille, Lille
  - Hôpital de la Croix Rousse, Lyon
  - Hopital La Pitie Salpetriere, Paris
  - Hopital Paul Brousse, Villejuif
- University of Zurich, Zurich, Switzerland
- United Kingdom (11):
  - Brighton & Sussex University Hospitals NHS Trust, Brighton
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Royal Liverpool & Broadgreen University Hospitals NHS Trust, Liverpool
  - Barts Health NHS Trust, London
  - Chelsea and Westminster Hospital, London
  - Imperial College, London
  - Kings College Hospital NHS Trust, London
  - Freeman Hospital, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital, Plymouth
  - Portsmouth Hospitals NHS Trust, Portsmouth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and North America. The first participant was screened on 01 September 2016. The last study visit occurred on 31 May 2018.
Pre-assignment Details: 166 participants were screened.
Groups:
- Selonsertib + Prednisolone: Participants received selonsertib (GS-4997) 18 mg tablet orally once daily + prednisolone 40 mg (4 x 10 mg tablets) orally once daily for 28 days.
- Placebo + Prednisolone: Participants received placebo-to-match selonsertib 18 mg tablet orally once daily + prednisolone 40 mg (4 x 10 mg tablets) orally once daily for 28 days.
Period: Overall Study
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Started | 52 | 52
Completed | 26 | 37
Not Completed | 26 | 15
Not completed — Adverse Event | 1 | 2
Not completed — Withdrew Consent | 3 | 2
Not completed — Investigator's Discretion | 2 | 0
Not completed — Death | 12 | 8
Not completed — Liver Biopsy Inconsistent With Diagnosis | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Subjects Randomized but Never Treated | 2 | 0
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who were randomized and took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (10.0) | 49 (9.3) | 49 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 29 | 36 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 46 | 49 | 95
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 44 | 44 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Hospitalized at Time of Screening [Count of Participants; unit: Participants]
  Yes | 46 | 48 | 94
  No | 4 | 4 | 8
Days Hospitalized Prior to First Dose Date [Mean (Standard Deviation); unit: Days] — Population: Only participants who were hospitalized were analyzed.
  Days
    number analyzed (Participants) | 46 | 48 | 94
    (all) | 10 (4.6) | 10 (5.2) | 10 (4.9)
Baseline Infection [Count of Participants; unit: Participants]
  Yes | 6 | 11 | 17
  No | 44 | 41 | 85
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: Units per liter (U/L)] — Population: Participants with available baseline values were analyzed.
  Units per liter (U/L)
    number analyzed (Participants) | 49 | 52 | 101
    (all) | 45 (33.5) | 48 (23.2) | 46 (28.5)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: U/L] — Population: Participants with available baseline values were analyzed.
  U/L
    number analyzed (Participants) | 49 | 52 | 101
    (all) | 122 (60.9) | 129 (59.9) | 126 (60.2)
Gamma Glutamyl Transferase (GGT) [Mean (Standard Deviation); unit: U/L] — Population: Participants with available baseline values were analyzed.
  U/L
    number analyzed (Participants) | 30 | 33 | 63
    (all) | 238 (175.5) | 278 (358.7) | 259 (285.0)
Alkaline Phosphatase [Mean (Standard Deviation); unit: U/L] — Population: Participants with available baseline values were analyzed.
  U/L
    number analyzed (Participants) | 49 | 52 | 101
    (all) | 162 (62.2) | 189 (111.3) | 176 (91.4)
Bilirubin [Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)] — Population: Participants with available baseline values were analyzed.
  Milligrams per deciliter (mg/dL)
    number analyzed (Participants) | 49 | 52 | 101
    (all) | 14.3 (8.35) | 14.5 (7.78) | 14.4 (8.02)
Albumin [Mean (Standard Deviation); unit: Grams per deciltre (g/dL)] — Population: Participants with available baseline values were analyzed.
  Grams per deciltre (g/dL)
    number analyzed (Participants) | 49 | 52 | 101
    (all) | 3.1 (0.62) | 3.0 (0.53) | 3.0 (0.58)
International Normalized Ratio (INR) [Mean (Standard Deviation); unit: Ratio] — Population: Participants with available baseline values were analyzed.
  Ratio
    number analyzed (Participants) | 47 | 52 | 99
    (all) | 1.7 (0.31) | 1.6 (0.22) | 1.6 (0.27)
Model for End-Stage Liver Disease (MELD) Score [Mean (Standard Deviation); unit: Units on a scale] — MELD scores are used to assess prognosis and suitability for liver transplantation. Scores can range from 6 to 40, with higher scores indicating greater disease severity.
  Units on a scale | 22 (4.2) | 22 (4.4) | 22 (4.3)
Child-Pugh-Turcotte (CPT) Score [Mean (Standard Deviation); unit: Units on a scale] — CPT scores are used to assess the severity of cirrhosis. Scores can range from 5 to 15, with higher scores indicating a greater severity of disease. Population: Participants with available baseline values were analyzed.
  Units on a scale
    number analyzed (Participants) | 47 | 52 | 99
    (all) | 10 (1.2) | 10 (1.3) | 10 (1.2)
Maddrey Discriminant Function (DF) Score [Mean (Standard Deviation); unit: Units on a scale] — Baseline Maddrey Discriminant Function (DF) score is a prognostic tool used to determine the next step of treatment based on the severity of AH. Maddrey DF score of < 32 indicates mild to moderate AH and a lower chance of death in the next few months. Maddrey DF score of ≥ 32 indicates severe AH and a higher chance of death in the next few months. The score has no bounds. Population: Participants with available baseline values were analyzed.
  Units on a scale
    number analyzed (Participants) | 44 | 52 | 96
    (all) | 42 (16.9) | 38 (11.4) | 40 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent (TE) Adverse Events (AE), Serious AEs (SAE), AEs Leading to Premature Study Drug Discontinuation, and Grade 3 or 4 Laboratory Abnormalities
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Laboratory toxicity grading was based on Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.
Time Frame: Up to Day 28 plus 30 days
Population: Safety Analysis Set included participants who were randomized and took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 50 | 52
Percentage of participants
  TEAEs | 94.0 | 94.2
  TE SAEs | 50.0 | 40.4
  TEAEs (discontinuation of Selonsertib/Placebo) | 18.0 | 7.7
  TEAEs (discontinuation of Prednisolone) | 14.0 | 11.5
  TEAEs (discontinuation of both drugs in regimen) | 14.0 | 7.7
  Laboratory abnormalities (Grade 3 or 4) | 72.0 | 72.0
  Laboratory abnormalities (Grade 3) | 42.0 | 52.0
  Laboratory abnormalities (Grade 4) | 30.0 | 20.0

2. Secondary Outcome: Percentage of Participants Who Died by Day 28
Description: The percentage of participants who died by Day 28 was calculated.
Time Frame: Day 28
Population: Participants in the Full Analysis Set (participants who took at least 1 dose of study drug, and had histologically-confirmed severe alcoholic hepatitis (AH)) with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 47 | 50
Percentage of participants | 4.3 | 4.0
Statistical Analysis 1: Comparison: Selonsertib + Prednisolone vs Placebo + Prednisolone; Test type: Superiority; p = 1.00, Fisher Exact; P-value from 2-sided Fisher's exact test was used to explore differences between treatment groups in the percentage of participants with an event

3. Secondary Outcome: Percentage of Participants Who Died by Week 8
Description: The percentage of participants who died by Week 8 was calculated.
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 44 | 49
Percentage of participants | 20.5 | 6.1
Statistical Analysis 1: Comparison: Selonsertib + Prednisolone vs Placebo + Prednisolone; Test type: Superiority; p = 0.061, Fisher Exact; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants Who Died by Week 12
Description: The percentage of participants who died by Week 12 was calculated.
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 43 | 49
Percentage of participants | 25.6 | 10.2
Statistical Analysis 1: Comparison: Selonsertib + Prednisolone vs Placebo + Prednisolone; Test type: Superiority; p = 0.060, Fisher Exact; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Died by Week 24
Description: The percentage of participants who died by Week 24 was calculated.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 41 | 48
Percentage of participants | 31.7 | 18.8
Statistical Analysis 1: Comparison: Selonsertib + Prednisolone vs Placebo + Prednisolone; Test type: Superiority; p = 0.22, Fisher Exact — P-value from 2-sided Fisher's exact test was used to explore differences between treatment groups in the percentage of participants with an event

6. Secondary Outcome: Percentage of Participants With Survival at Day 28 Using Kaplan-Meier
Description: The percentage of participants with survival at Day 28 using Kaplan-Meier was calculated.
Time Frame: Day 28
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 51
Percentage of participants | 95.7 [84.0 to 98.9] | 96.1 [85.2 to 99.0]

7. Secondary Outcome: Percentage of Participants With Survival at Week 8 Using Kaplan-Meier
Description: The percentage of participants with survival at Week 8 using Kaplan-Meier was calculated.
Time Frame: Week 8
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 51
Percentage of participants | 80.0 [65.1 to 89.1] | 94.0 [82.6 to 98.0]

8. Secondary Outcome: Percentage of Participants With Survival at Week 12 Using Kaplan-Meier
Description: The percentage of participants with survival at Week 12 using Kaplan-Meier was calculated.
Time Frame: Week 12
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 51
Percentage of participants | 75.3 [59.8 to 85.5] | 89.9 [77.5 to 95.7]

9. Secondary Outcome: Percentage of Participants With Survival at Week 24 Using Kaplan-Meier
Description: The percentage of participants with survival at Week 24 using Kaplan-Meier was calculated.
Time Frame: Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 51
Percentage of participants | 70.3 [54.3 to 81.6] | 81.7 [67.7 to 90.0]

10. Secondary Outcome: Percentage of Participants Who Received a Liver Transplant
Description: The percentage of participants who received a liver transplant by week 24 was calculated.
Time Frame: Day 28, Week 8, Week 12, and Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 45 | 48
Percentage of participants
  Day 28 | 2.2 | 0
  Week 8: number analyzed (Participants) | 36 | 46
  Week 8 | 2.8 | 0
  Week 12: number analyzed (Participants) | 33 | 44
  Week 12 | 3.0 | 0
  Week 24: number analyzed (Participants) | 29 | 39
  Week 24 | 6.9 | 2.6

11. Secondary Outcome: Percentage of Participants With Hepatorenal Syndrome (HRS)
Description: The occurrence of HRS was confirmed based on the following diagnostic criteria from the International Ascites Club (IAC): 1) Cirrhosis with ascites, 2) Diagnosis of acute kidney injury (AKI) according to the ICA-AKI criteria, 3) Absence of shock, 4) No current or recent treatment with nephrotoxic drugs, and 5) Absence of parenchymal renal disease as indicated by proteinuria >500 mg/day, microhematuria (> 50 red blood cells per high power field) and/or abnormal renal ultrasonography.
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 51
Percentage of participants | 4.2 | 2.0

12. Secondary Outcome: Percentage of Participants With Infection
Description: The occurrence of bacterial, fungal, or viral infections was recorded. An infection was considered definite in participants with clinical evidence of infection and a positive culture from a normally sterile source (with the exception of spontaneous bacterial peritonitis).
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 51
Percentage of participants | 37.5 | 29.4

13. Secondary Outcome: Length of Hospital Stay
Description: Length of initial hospital stay from first dose date of study drug was calculated for participants who were released from initial hospitalization separately from those who died during their initial hospitalization.
Time Frame: Up to 24 weeks
Population: Participants in the Full Analysis Set with available data were analyzed. Participants released from initial hospitalization and those who died during initial hospitalization were analyzed separately, so a total of 41 participants and 45 participants were analyzed for the Selonsertib + Prednisolone and Placebo + Prednisolone arms, respectively.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 41 | 45
Days
  Released from initial hospitalization: number analyzed (Participants) | 38 | 43
  Released from initial hospitalization | 11.0 (11.53) | 11.0 (11.25)
  Died during initial hospitalization: number analyzed (Participants) | 3 | 2
  Died during initial hospitalization | 36.0 (18.52) | 6.0 (1.41)

14. Secondary Outcome: Change From Baseline in Liver Biochemistry Tests: Alanine Aminotransferase (ALT)
Description: Change from Baseline was calculated as the value at endpoint minus the value at Baseline.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 47 | 49
U/L
  Change at Week 1: number analyzed (Participants) | 45 | 47
  Change at Week 1 | 26 (40.7) | 29 (28.2)
  Change at Week 2: number analyzed (Participants) | 42 | 46
  Change at Week 2 | 31 (35.0) | 36 (33.6)
  Change at Week 3: number analyzed (Participants) | 39 | 46
  Change at Week 3 | 24 (32.6) | 24 (28.8)
  Change at Week 4: number analyzed (Participants) | 35 | 46
  Change at Week 4 | 15 (28.7) | 12 (32.6)
  Change at Week 6: number analyzed (Participants) | 32 | 40
  Change at Week 6 | -10 (19.9) | -18 (21.8)
  Change at Week 8: number analyzed (Participants) | 30 | 42
  Change at Week 8 | -13 (18.1) | -20 (24.6)
  Change at Week 12: number analyzed (Participants) | 27 | 39
  Change at Week 12 | -15 (19.3) | -17 (42.9)
  Change at Week 16: number analyzed (Participants) | 28 | 36
  Change at Week 16 | -14 (21.0) | -21 (28.6)
  Change at Week 20: number analyzed (Participants) | 24 | 35
  Change at Week 20 | -12 (18.6) | -24 (21.7)
  Change at Week 24: number analyzed (Participants) | 25 | 35
  Change at Week 24 | -12 (19.4) | -22 (21.8)

15. Secondary Outcome: Change From Baseline in Liver Biochemistry Tests: Aspartate Aminotransferase (AST)
Description: Change from Baseline was calculated as the value at endpoint minus the value at Baseline.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 47 | 49
U/L
  Change at Week 1: number analyzed (Participants) | 45 | 45
  Change at Week 1 | -2 (66.9) | 4 (52.8)
  Change at Week 2: number analyzed (Participants) | 40 | 43
  Change at Week 2 | -17 (58.5) | -11 (52.9)
  Change at Week 3: number analyzed (Participants) | 39 | 45
  Change at Week 3 | -34 (38.4) | -39 (54.0)
  Change at Week 4: number analyzed (Participants) | 35 | 44
  Change at Week 4 | -45 (35.8) | -55 (60.2)
  Change at Week 6: number analyzed (Participants) | 32 | 40
  Change at Week 6 | -54 (45.6) | -74 (60.0)
  Change at Week 8: number analyzed (Participants) | 30 | 42
  Change at Week 8 | -48 (46.6) | -61 (63.5)
  Change at Week 12: number analyzed (Participants) | 27 | 37
  Change at Week 12 | -59 (45.2) | -63 (86.5)
  Change at Week 16: number analyzed (Participants) | 26 | 36
  Change at Week 16 | -59 (56.9) | -70 (76.4)
  Change at Week 20: number analyzed (Participants) | 24 | 35
  Change at Week 20 | -57 (46.9) | -64 (72.6)
  Change at Week 24: number analyzed (Participants) | 25 | 35
  Change at Week 24 | -59 (49.6) | -68 (59.4)

16. Secondary Outcome: Change From Baseline in Liver Biochemistry Tests: Gamma Glutamyl Transferase (GGT)
Description: Change from Baseline was calculated as the value at endpoint minus the value at Baseline.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 29 | 33
U/L
  Change at Week 1: number analyzed (Participants) | 26 | 31
  Change at Week 1 | 3 (79.2) | -1 (192.5)
  Change at Week 2: number analyzed (Participants) | 26 | 31
  Change at Week 2 | 9 (140.8) | 9 (189.0)
  Change at Week 3: number analyzed (Participants) | 24 | 32
  Change at Week 3 | -12 (170.2) | 9 (197.1)
  Change at Week 4: number analyzed (Participants) | 25 | 30
  Change at Week 4 | -7 (169.3) | -5 (284.0)
  Change at Week 6: number analyzed (Participants) | 22 | 26
  Change at Week 6 | -61 (139.7) | -72 (173.4)
  Change at Week 8: number analyzed (Participants) | 22 | 29
  Change at Week 8 | -96 (137.7) | -121 (314.2)
  Change at Week 12: number analyzed (Participants) | 20 | 26
  Change at Week 12 | -105 (136.1) | -100 (274.0)
  Change at Week 16: number analyzed (Participants) | 20 | 23
  Change at Week 16 | -87 (157.4) | -114 (251.3)
  Change at Week 20: number analyzed (Participants) | 18 | 24
  Change at Week 20 | -134 (150.9) | -85 (342.9)
  Change at Week 24: number analyzed (Participants) | 20 | 25
  Change at Week 24 | -131 (154.4) | -54 (277.0)

17. Secondary Outcome: Change From Baseline in Liver Biochemistry Tests: Alkaline Phosphatase
Description: Change from Baseline was calculated as the value at endpoint minus the value at Baseline.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 47 | 49
U/L
  Change at Week 1: number analyzed (Participants) | 45 | 47
  Change at Week 1 | 11 (55.3) | -3 (63.6)
  Change at Week 2: number analyzed (Participants) | 42 | 46
  Change at Week 2 | 23 (70.7) | -5 (70.6)
  Change at Week 3: number analyzed (Participants) | 39 | 46
  Change at Week 3 | 10 (68.7) | -4 (89.8)
  Change at Week 4: number analyzed (Participants) | 35 | 46
  Change at Week 4 | 8 (71.7) | -16 (89.8)
  Change at Week 6: number analyzed (Participants) | 34 | 40
  Change at Week 6 | 1 (65.3) | -21 (69.8)
  Change at Week 8: number analyzed (Participants) | 30 | 42
  Change at Week 8 | -14 (52.6) | -47 (97.8)
  Change at Week 12: number analyzed (Participants) | 27 | 40
  Change at Week 12 | -35 (65.0) | -52 (102.8)
  Change at Week 16: number analyzed (Participants) | 28 | 36
  Change at Week 16 | -26 (83.1) | -50 (92.8)
  Change at Week 20: number analyzed (Participants) | 24 | 35
  Change at Week 20 | -29 (83.3) | -45 (106.8)
  Change at Week 24: number analyzed (Participants) | 25 | 36
  Change at Week 24 | -25 (87.3) | -43 (101.0)

18. Secondary Outcome: Change From Baseline in Liver Biochemistry Tests: Bilirubin
Description: Change from Baseline was calculated as the value at endpoint minus the value at Baseline.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 47 | 49
mg/dL
  Change at Week 1: number analyzed (Participants) | 44 | 47
  Change at Week 1 | -2.1 (3.99) | -4.3 (3.46)
  Change at Week 2: number analyzed (Participants) | 42 | 46
  Change at Week 2 | -2.9 (5.34) | -6.3 (4.99)
  Change at Week 3: number analyzed (Participants) | 39 | 46
  Change at Week 3 | -4.8 (7.68) | -7.2 (6.21)
  Change at Week 4: number analyzed (Participants) | 35 | 46
  Change at Week 4 | -6.3 (6.01) | -8.6 (6.52)
  Change at Week 6: number analyzed (Participants) | 32 | 40
  Change at Week 6 | -8.7 (8.22) | -9.3 (7.40)
  Change at Week 8: number analyzed (Participants) | 30 | 42
  Change at Week 8 | -8.4 (7.53) | -10.3 (7.36)
  Change at Week 12: number analyzed (Participants) | 27 | 40
  Change at Week 12 | -9.5 (7.86) | -11.2 (7.79)
  Change at Week 16: number analyzed (Participants) | 28 | 36
  Change at Week 16 | -9.4 (8.35) | -11.3 (8.37)
  Change at Week 20: number analyzed (Participants) | 24 | 35
  Change at Week 20 | -8.1 (9.88) | -11.3 (7.94)
  Change at Week 24: number analyzed (Participants) | 25 | 36
  Change at Week 24 | -9.4 (7.72) | -10.7 (8.09)

19. Secondary Outcome: Change From Baseline in Liver Biochemistry Tests: Albumin
Description: Change from Baseline was calculated as the value at endpoint minus the value at Baseline.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 47 | 49
g/dL
  Change at Week 1: number analyzed (Participants) | 45 | 47
  Change at Week 1 | 0.2 (0.45) | 0.2 (0.31)
  Change at Week 2: number analyzed (Participants) | 42 | 46
  Change at Week 2 | 0.3 (0.47) | 0.4 (0.45)
  Change at Week 3: number analyzed (Participants) | 39 | 46
  Change at Week 3 | 0.3 (0.58) | 0.4 (0.54)
  Change at Week 4: number analyzed (Participants) | 35 | 46
  Change at Week 4 | 0.4 (0.63) | 0.5 (0.57)
  Change at Week 6: number analyzed (Participants) | 34 | 40
  Change at Week 6 | 0.2 (0.82) | 0.4 (0.67)
  Change at Week 8: number analyzed (Participants) | 30 | 42
  Change at Week 8 | 0.3 (0.80) | 0.6 (0.66)
  Change at Week 12: number analyzed (Participants) | 27 | 40
  Change at Week 12 | 0.5 (0.82) | 0.6 (0.68)
  Change at Week 16: number analyzed (Participants) | 28 | 36
  Change at Week 16 | 0.5 (0.95) | 0.7 (0.64)
  Change at Week 20: number analyzed (Participants) | 24 | 35
  Change at Week 20 | 0.8 (0.92) | 0.8 (0.68)
  Change at Week 24: number analyzed (Participants) | 25 | 36
  Change at Week 24 | 0.8 (0.76) | 0.8 (0.68)

20. Secondary Outcome: Change From Baseline in Liver Biochemistry Tests: International Normalized Ratio (INR)
Description: Change from Baseline was calculated as the value at endpoint minus the value at Baseline.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 45 | 49
Ratio
  Change at Week 1: number analyzed (Participants) | 42 | 47
  Change at Week 1 | -0.1 (0.28) | -0.1 (0.16)
  Change at Week 2: number analyzed (Participants) | 39 | 45
  Change at Week 2 | -0.2 (0.32) | -0.2 (0.23)
  Change at Week 3: number analyzed (Participants) | 34 | 43
  Change at Week 3 | -0.3 (0.38) | -0.2 (0.25)
  Change at Week 4: number analyzed (Participants) | 33 | 46
  Change at Week 4 | -0.3 (0.36) | -0.2 (0.18)
  Change at Week 6: number analyzed (Participants) | 31 | 40
  Change at Week 6 | -0.2 (0.40) | -0.2 (0.33)
  Change at Week 8: number analyzed (Participants) | 26 | 42
  Change at Week 8 | -0.3 (0.43) | -0.3 (0.19)
  Change at Week 12: number analyzed (Participants) | 23 | 40
  Change at Week 12 | -0.3 (0.41) | -0.3 (0.19)
  Change at Week 16: number analyzed (Participants) | 26 | 35
  Change at Week 16 | -0.3 (0.40) | -0.3 (0.22)
  Change at Week 20: number analyzed (Participants) | 22 | 34
  Change at Week 20 | -0.3 (0.42) | -0.3 (0.27)
  Change at Week 24: number analyzed (Participants) | 25 | 34
  Change at Week 24 | -0.4 (0.36) | -0.3 (0.32)

21. Secondary Outcome: Percentage of Participants With Lille Response (Score < 0.45) at Day 7
Description: The Lille score is a tool used to predict which participants with severe alcoholic hepatitis (AH) were not responding to corticosteroid therapy. It ranges between 0 and 1, with low scores (< 0.16) indicating complete response or positive response to steroids (continue therapy) and high scores (≥ 0.56) indicating no response or poor response to steroids (stop therapy). The Lille score was calculated using baseline factors: age, albumin, total bilirubin, serum creatinine, prothrombin time; and the change in total bilirubin between baseline (Day 1) and Day 7. Lille response was defined as having a Lille score < 0.45.
Time Frame: Day 7
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 51
Percentage of participants | 77.1 | 86.3
Statistical Analysis 1: Comparison: Selonsertib + Prednisolone vs Placebo + Prednisolone; Test type: Superiority; p = 0.30, Fisher Exact; Fisher's exact test (2-sided) was used to explore differences between groups in the percentage of participants with response/non-response

22. Secondary Outcome: Percentage of Participants With a Lille Null Response (Score ≥ 0.56) at Day 7
Description: The Lille score is a tool used to predict which participants with severe AH were not responding to corticosteroid therapy. It ranges between 0 and 1, with low scores (< 0.16) indicating complete response or positive response to steroids (continue therapy) and high scores (≥ 0.56) indicating no response or poor response to steroids (stop therapy). The Lille score was calculated using baseline factors: age, albumin, total bilirubin, serum creatinine, prothrombin time; and the change in total bilirubin between baseline (Day 1) and Day 7. Lille null response was defined as having a Lille score ≥ 0.56.
Time Frame: Day 7
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 51
Percentage of participants | 14.6 | 7.8

23. Secondary Outcome: Lille Score at Day 7 as a Continuous Variable
Description: The Lille score is a tool used to predict which participants with severe AH were not responding to corticosteroid therapy. It ranges between 0 and 1, with low scores (< 0.16) indicating complete response or positive response to steroids (continue therapy) and high scores (≥ 0.56) indicating no response or poor response to steroids (stop therapy). The Lille score was calculated using baseline factors: age, albumin, total bilirubin, serum creatinine, prothrombin time; and the change in total bilirubin between baseline (Day 1) and Day 7.
Time Frame: Day 7
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Lille score
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 47 | 48
Lille score | 0.254 (0.2495) | 0.178 (0.1534)

24. Secondary Outcome: Percentage of Participants With Estimated Mortality at Month 2 and Month 6: Combined Scoring Including Lille Score at Day 7 and Baseline Model for End-Stage Liver Disease (MELD) Score
Description: The Lille score is a tool used to predict which participants with severe AH were not responding to corticosteroid therapy. It ranges between 0 and 1, with low scores (< 0.16) indicating complete response or positive response to steroids (continue therapy) and high scores (≥ 0.56) indicating no response or poor response to steroids (stop therapy). MELD scores are used to assess prognosis and suitability for liver transplantation. Scores can range from 6 to 40, with higher scores indicating greater disease severity. A scoring system combining the Lille score at Day 7 and the baseline MELD score was used to calculate the percentage of participants expected to die by Month 2 and by Month 6.
Time Frame: Baseline and Day 7 Time Points used to calculate Overall Mortality Risk at Months 2 and 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 47 | 48
Percentage of participants
  Mortality Risk at Month 2 | 13.0 (10.94) | 9.7 (6.57)
  Mortality Risk at Month 6 | 19.8 (15.15) | 15.2 (9.28)

25. Secondary Outcome: Change From Baseline in Prognostic Index: Model for End-Stage Liver Disease (MELD) Score
Description: MELD scores are used to assess prognosis and suitability for liver transplantation. Scores can range from 6 to 40, with higher scores indicating greater disease severity. Change from Baseline was calculated as the value at endpoint minus the value at Baseline.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 48 | 49
Units on a scale
  Change at Week 1: number analyzed (Participants) | 44 | 47
  Change at Week 1 | -2 (2.9) | -3 (2.6)
  Change at Week 2: number analyzed (Participants) | 42 | 45
  Change at Week 2 | -3 (4.0) | -5 (3.5)
  Change at Week 3: number analyzed (Participants) | 36 | 43
  Change at Week 3 | -4 (4.7) | -5 (3.9)
  Change at Week 4: number analyzed (Participants) | 35 | 46
  Change at Week 4 | -5 (5.2) | -6 (3.9)
  Change at Week 6: number analyzed (Participants) | 32 | 39
  Change at Week 6 | -6 (6.1) | -7 (5.2)
  Change at Week 8: number analyzed (Participants) | 28 | 41
  Change at Week 8 | -7 (5.9) | -8 (4.7)
  Change at Week 12: number analyzed (Participants) | 26 | 40
  Change at Week 12 | -7 (6.0) | -10 (4.8)
  Change at Week 16: number analyzed (Participants) | 29 | 35
  Change at Week 16 | -7 (6.5) | -9 (5.5)
  Change at Week 20: number analyzed (Participants) | 23 | 34
  Change at Week 20 | -8 (7.6) | -10 (5.4)
  Change at Week 24: number analyzed (Participants) | 26 | 34
  Change at Week 24 | -9 (6.1) | -10 (5.6)

26. Secondary Outcome: Change From Baseline in Prognostic Index: Child-Pugh-Turcotte (CPT) Score
Description: CPT scores are used to assess the severity of cirrhosis. Scores can range from 5 to 15, with higher scores indicating a greater severity of disease
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 45 | 49
Units on a scale
  Change at Week 1: number analyzed (Participants) | 41 | 47
  Change at Week 1 | 0 (1.5) | -1 (0.9)
  Change at Week 2: number analyzed (Participants) | 39 | 45
  Change at Week 2 | -1 (1.4) | -1 (1.4)
  Change at Week 3: number analyzed (Participants) | 34 | 43
  Change at Week 3 | -1 (1.7) | -1 (1.4)
  Change at Week 4: number analyzed (Participants) | 33 | 46
  Change at Week 4 | -1 (1.9) | -2 (1.7)
  Change at Week 6: number analyzed (Participants) | 28 | 39
  Change at Week 6 | -1 (2.1) | -2 (1.7)
  Change at Week 8: number analyzed (Participants) | 26 | 41
  Change at Week 8 | -2 (2.4) | -2 (1.5)
  Change at Week 12: number analyzed (Participants) | 23 | 40
  Change at Week 12 | -2 (2.2) | -3 (1.7)
  Change at Week 16: number analyzed (Participants) | 26 | 35
  Change at Week 16 | -2 (2.4) | -3 (1.8)
  Change at Week 20: number analyzed (Participants) | 22 | 34
  Change at Week 20 | -3 (2.3) | -3 (1.6)
  Change at Week 24: number analyzed (Participants) | 24 | 34
  Change at Week 24 | -3 (1.7) | -3 (1.6)

27. Secondary Outcome: Change From Baseline in Prognostic Index: Maddrey Discriminant Function (DF) Score
Description: Baseline Maddrey DF score is a prognostic tool used to determine the next step of treatment based on the severity of AH. Maddrey DF score of < 32 indicates mild to moderate AH and a lower chance of death in the next few months. Maddrey DF score of ≥ 32 indicates severe AH and a higher chance of death in the next few months. The score has no bounds.
Time Frame: Baseline (Day 1) and up to 24 weeks
Population: Participants in the Full Analysis Set with available baseline and any postbaseline data were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
Number analyzed (Participants) | 42 | 49
Units on a scale
  Change at Week 1: number analyzed (Participants) | 39 | 47
  Change at Week 1 | -8 (15.2) | -10 (7.7)
  Change at Week 2: number analyzed (Participants) | 37 | 45
  Change at Week 2 | -13 (18.1) | -15 (11.4)
  Change at Week 3: number analyzed (Participants) | 33 | 43
  Change at Week 3 | -17 (21.8) | -17 (13.3)
  Change at Week 4: number analyzed (Participants) | 31 | 46
  Change at Week 4 | -19 (20.0) | -19 (10.9)
  Change at Week 6: number analyzed (Participants) | 27 | 39
  Change at Week 6 | -20 (23.2) | -19 (17.6)
  Change at Week 8: number analyzed (Participants) | 25 | 41
  Change at Week 8 | -19 (21.5) | -21 (12.0)
  Change at Week 12: number analyzed (Participants) | 22 | 40
  Change at Week 12 | -23 (21.8) | -23 (12.2)
  Change at Week 16: number analyzed (Participants) | 24 | 35
  Change at Week 16 | -23 (22.6) | -23 (13.7)
  Change at Week 20: number analyzed (Participants) | 21 | 34
  Change at Week 20 | -25 (26.2) | -23 (15.4)
  Change at Week 24: number analyzed (Participants) | 23 | 34
  Change at Week 24 | -27 (21.7) | -22 (16.9)

ADVERSE EVENTS:
Time Frame: Adverse Events: Up to Day 28 plus 30 days; All-Cause Mortality: Up to 24 weeks
Description: Safety Analysis Set included all participants who were randomized and took at least 1 dose of study drug.
Arm/Group | Selonsertib + Prednisolone | Placebo + Prednisolone
All-Cause Mortality (participants affected / at risk) | 14/50 | 9/52
Serious Adverse Events (participants affected / at risk) | 25/50 | 21/52
Other Adverse Events (participants affected / at risk) | 43/50 | 42/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selonsertib + Prednisolone (N=50) | Placebo + Prednisolone (N=52)
Coagulopathy (Blood and lymphatic system disorders) | 3 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 2
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 2 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0
Fungal abscess central nervous system (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2
Pneumonia legionella (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Uterine infection (Infections and infestations) | 0 | 1
Wound infection fungal (Infections and infestations) | 1 | 0
Blood lactic acid increased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coma hepatic (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 2 | 5
Confusional state (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selonsertib + Prednisolone (N=50) | Placebo + Prednisolone (N=52)
Leukocytosis (Blood and lymphatic system disorders) | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Ascites (Gastrointestinal disorders) | 15 | 14
Constipation (Gastrointestinal disorders) | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 6 | 2
Varices oesophageal (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 4 | 2
Fatigue (General disorders) | 4 | 6
Oedema (General disorders) | 4 | 6
Oedema peripheral (General disorders) | 12 | 11
Pyrexia (General disorders) | 1 | 4
Escherichia urinary tract infection (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 4
Headache (Nervous system disorders) | 1 | 3
Hepatic encephalopathy (Nervous system disorders) | 12 | 7
Agitation (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 5 | 5
Acute kidney injury (Renal and urinary disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Hypotension (Vascular disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Study Protocol: Original (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT02854631/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT02854631/Prot_001.pdf
  • Study Protocol: Amendment 2 (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02854631/Prot_002.pdf
  • Study Protocol: Amendment 3 (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT02854631/Prot_003.pdf
  • Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02854631/SAP_004.pdf